CLINICAL TRIAL: NCT01038492
Title: Testing the Feasibility of Using an Epigenetic Marker, p16, to Promote Smoking Cessation
Brief Title: p16 Methylation for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Durham VA Medical Center (U.S. Federal Agency); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00012350; 155923 (Other Grant/Funding Number: Cancer and Lymphoma Study Group B); 01344 (Other: Durham VAMC)
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2012-03

CONDITIONS: Tobacco Use Disorder; Smoking Cessation; Lung Cancer
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- p16 Methylation in Sputum Testing (Experimental): * Patients tested for smoking-related changes in their breathing
  * shown a presentation on development of lung cancer
  * complete a questionnaire on items from presentation, desire to have p16 methylation test, views regarding their health and lung cancer, current smoking habits, and demographic detail
  * given a sputum cup which they are asked to spit into on three consecutive mornings and then return to the lab for processing
  * a results letter is mailed to them and then followed up with a phone call at one month to discuss the results as well as any changes in their attitudes or smoking habits
  * patients are called again at three months and asked about any changes in their attitudes or smoking habits
  Interventions: Behavioral: p16 Methylation and Lung Cancer Education

INTERVENTIONS:
Behavioral: p16 Methylation and Lung Cancer Education — * patients shown a presentation on p16 methylation and the development of lung cancer, asked to complete a questionnaire on items from presentation, desire to have p16 methylation test, views regarding their health and lung cancer, current smoking habits, and demographic details
  * patients given a sputum cup which they are asked to spit into on three consecutive mornings and then return to the lab for processing
  * a results letter is mailed to them and then followed up with a phone call at one month to discuss the results as well as any changes in their attitudes or smoking habits
  * patients are called again at three months and asked about any changes in their attitudes or smoking habits.
  Other Names: Lung cancer education

SUMMARY:
Smoking cessation is often difficult for smokers to achieve for a variety of reasons including: difficulty with nicotine withdrawal, failure to perceive the benefits of smoking cessation, and failure to perceive the risks associated with smoking. We argue that the most effective biomarkers to affect perceptions of harm, especially for lung cancer, are those that signal progression towards disease development Proposed is a pilot study of educating smokers about the role of genetics and lung cancer in Durham VA out-patient clinics. The goal of this pilot study is to assess the interest in study participation from the VA smoking population, as well as to determine the fraction of subjects who will complete the study to power a future larger trial. Interested patients will receive a 15 minute educational presentation on the function of p16 and its role in development of lung cancer. They will then be assessed for airway obstruction by hand-held spirometry followed by review of a questionnaire assessing their understanding of the presented information, their concern for developing lung cancer, and their desire to quit smoking. All patients will be offered smoking cessation assistance at this point. Enrolled patients will then be given 3 sputum cups to take home and return with morning sputum samples by mail. Samples will be assessed for evidence of p16 methylation and patients will be informed of the results. Follow-up phone interviews will be performed at 2 to 4 weeks after patients have received their results by mail to assess their understanding of the results, and their desire to stop smoking. A final phone interview will occur approximately 3 months after the sputum testing to assess attempts to stop smoking as well as the patients continued understanding of their test results. For purposes of this pilot, we are interested primarily in the descriptive statistics (e.g., frequencies) associated with the outcome of each objective (e.g., how many expressed interest, how many returned the sputum samples).

DETAILED DESCRIPTION:
In the United States during 2007, ~ 213,380 people were expected to be diagnosed with lung cancer, and ~ 160,390 expected to die of the disease. Among those diagnosed with lung cancer, 79% to 90% are cigarette smokers. Overall, ~21% of adults in the U.S. smoke. The most important and cost-effective strategy for the prevention of lung cancer mortality is smoking avoidance and cessation. Smoking cessation is often difficult for smokers to achieve for a variety of reasons including: difficulty with nicotine withdrawal, failure to perceive the benefits of smoking cessation, and failure to perceive the risks associated with smoking. We argue that the most effective biomarkers to affect perceptions of harm, especially for lung cancer, are those that signal progression towards disease development. Prior to the development of lung cancer, there are genetic alterations in the bronchial epithelium. One such alteration is the methylation of the promoter region of Rb-p16 (p16) important in regulation of the G1-S transition of the cell cycle. Prior studies have shown that presence of the promoter methylation of p16 results in a 2-fold increase in risk of developing lung cancer in smokers with evidence of airway obstruction.

Proposed is a pilot study of educating smokers about the role of genetics and lung cancer in Durham VA out-patient clinics. The goal of this pilot study is to assess the interest in study participation from the VA smoking population, as well as to determine the fraction of subjects who will complete the study to power a future larger trial. Interested patients will receive a 15 minute educational presentation on the function of p16 and its role in development of lung cancer. They will then be assessed for airway obstruction by hand-held spirometry followed by review of a questionnaire assessing their understanding of the presented information, their concern for developing lung cancer, and their desire to quit smoking. All patients will be offered smoking cessation assistance at this point. Enrolled patients will then be given 3 sputum cups to take home and return with morning sputum samples by mail. Samples will be assessed for evidence of p16 methylation and patients will be informed of the results. Follow-up phone interviews will be performed at 2 to 4 weeks after patients have received their results by mail to assess their understanding of the results, and their desire to stop smoking. A final phone interview will occur approximately 3 months after the sputum testing to assess attempts to stop smoking as well as the patients continued understanding of their test results. Patients will be compensated a total of $40.00 for completing the study. For purposes of this pilot, we are interested primarily in the descriptive statistics (e.g., frequencies) associated with the outcome of each objective (e.g., how many expressed interest, how many returned the sputum samples).

ELIGIBILITY:
Inclusion Criteria:

* current smoker
* >30 pack year history
* FEV1/FVC<70%
* patients in outpatient pulmonary clinics at Durham VAMC and general medicine outpatient clinics at Durham VA Hillandale Clinic

Exclusion Criteria:

* diagnosis of head, neck, or lung cancer
* diagnosis of psychosis or severe cognitive impairment
* refusal to sign informed consent
* severe speech or hearing impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine patient interest in finding out whether, through the testing of p16 methylation in their sputum, whether they are at increased or average risk for developing cancer | 3 months
To determine the percentage of patients who return their sputum for p16 methylation analysis | 3 months
To determine the percentage of patients who complete the 1-month phone interview | 3 months
To determine the percentage of patients who complete the 3-month interview | 3 months

SECONDARY OUTCOMES:
To determine the percentage of patients who have a positive result for p16 methylation in their sputum, indicating they are at higher risk for developing lung cancer | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott Shofer, MD, PhD, Principal Investigator — Durham VA Medical Center/Duke University Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Shofer S, Beyea M, Li S, Bastian LA, Wahidi MM, Kelley M, Lipkus IM. Feasibility of using an epigenetic marker of risk for lung cancer, methylation of p16, to promote smoking cessation among US veterans. BMJ Open Respir Res. 2014 Jun 28;1(1):e000032. doi: 10.1136/bmjresp-2014-000032. eCollection 2014. PMID 25478181